CLINICAL TRIAL: NCT06174155
Title: Botulinum Toxin-A Injection and Shock Waves on Hypertrophic Scars in Hand-burned Children
Brief Title: Comparative Study Between Botulinum Toxin-A Injection and Shock Waves on Hypertrophic Scars in Hand-burned Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Saeed Alsakhawi, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004732
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Hand-burned Children
MeSH Terms: interventions — Physical Therapy Modalities; Botulinum Toxins, Type A; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): The control group will receive the physical therapy program and conduct five times per week over four consecutive weeks under the supervision of a physical rehabilitation specialist.
  Interventions: Other: physical therapy treatment
- Study group A (Active Comparator): The study group A will receive Botulinum toxin-A injection in addition to physical therapy program as control group
  Interventions: Other: Botulinum toxin-A injection in addition to physical therapy program
- Study group B (Active Comparator): The study group B will receive shock wave therapy in addition to physical therapy program as control group.
  Interventions: Other: shock wave therapy in addition to physical therapy program

INTERVENTIONS:
Other: physical therapy treatment — The control group will receive the physical therapy program and conduct five times per week over four consecutive weeks under the supervision of a physical rehabilitation specialist. The primary focus of the program was to improve scar malleability, lengthen muscles and tendons, enhance joint mobility, and to restore functionality. Each session lasted almost for 45 minutes and consisted of therapeutic paraffin application; deep tissue massaging (5 minutes); stretching exercises; active ROM exercises.
  Arms: Control group
Other: Botulinum toxin-A injection in addition to physical therapy program — Two injection procedures will be used. The first is an EMG-guided BTX-A administration (Botox®, Allergan PLC, Dublin, Ireland) that will be localized to the motor endplate zone of the wrist flexors, radial and ulnar deviators. The second is a meso-injection procedure, where the BTX-A will be injected subdermal, intradermal, and into the scar (around the periphery and into the center).
  Arms: Study group A
Other: shock wave therapy in addition to physical therapy program — After wound and skin graft healing (~ 90 days post-surgery), the unfocused shockwave will be applied to the site of burn injury on the volar aspect of the hand of the subjects and will allocate to the shock wave therapy intervention arm. The treatment will be delivered using a portable shockwave device (Zimmer enPuls, EMS physio Ltd, Germany).
  Arms: Study group B

SUMMARY:
PURPOSE: The study aims to compare study between Botulinum toxin-A injection and shock waves therapy on hypertrophic scars in hand-burned children.

BACKGROUND: Burn injuries can cause significant physical and psychological distress, especially when they result in hypertrophic scarring. In children, who are particularly vulnerable to these injuries, it is important to accurately assess the severity of these scars and their impact on functionality.

HYPOTHESES: There is no significant difference between the combined effect of the traditional physical therapy program with botulinum toxin-A injection and the traditional physical therapy program with shock waves therapy on improving wrist extension, ulnar deviation, radial deviation, hand grip strength, and severity of the scar on hypertrophic scars in hand-burned children.

ELIGIBILITY:
Inclusion Criteria:

* Age will range from 6-18 years
* Diagnosed with hypertrophic scars resulting from hand burns.
* Has burn injuries caused by flame, scald or chemical agents.
* With a total body surface area (TBSA) varied from 10 to 30%
* A resistant partial or complete loss of wrist flexion attributable to wrist flexor contracture
* After wound and skin graft healing (~ 90 days post-surgery),

Exclusion criteria:

* Children with underlying medical conditions that could interfere with scar healing or treatment outcomes
* Skin flap surgery, malignancies, cardiac arrhythmias, pacemaker implantation, coagulopathies, fractures about the treatment area, articular adhesions, and psychiatric co-morbidities

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Electronic goniometer | 3 months
  to assess the range of motions of wrist extension, radial deviation, and ulnar deviation. Active ROM Measurement: the patient independently moving their affected joint. The device records the joint angle throughout the movement, allowing for a thorough assessment of functional limitations caused by hypertrophic scars. Passive ROM Measurement: the therapist moves the patient's joint through its range of motion while the electronic goniometer measures and records the joint angles. This approach provides valuable information about the degree of movement restriction due to hypertrophic scarring.
Hand grip Dynamometer | 3 months
  for hand grip strength is used for assessing upper limb impairment, work capacity following injury or disease, and rehabilitation progression and/or potential following injury or surgery. For each child, the maximal voluntary contraction was determined as the highest of three contractions (INITIAL MAX). After a one-minute rest period, children will be instructed to squeeze the dynamometer in a static contraction at a level of 50% maximal for as long as possible, the duration of which will be recorded (DURATION). The level of static contraction will be monitored by the assessor who provided verbal feedback to ensure that a level of 50% maximal was maintained. Children must perform an additional post-fatigue maximal contraction within 10 seconds of completing the 50% maximal static contraction (FINAL MAX).
Vancouver scar scale | 3 months
  It employs four main parameters to evaluate hypertrophic scars: vascularity, pigmentation, pliability, and height. These parameters are individually scored on a scale ranging from 0 to 3, with higher scores indicating greater severity. The scores are then summed to provide an overall measure of scar severity, ranging from 0 (normal skin) to 14 (most severe scar). To ensure accurate evaluations, it is recommended to have adequate lighting, a calm environment, and reliable observers trained in using the VSS. Evaluators carefully assess each parameter, considering factors such as erythema, texture, and skin tension to assign appropriate scores. Finally, the total score provides a comprehensive representation of the hypertrophic scar's severity.

CONTACTS AND LOCATIONS:
Overall Officials: Reham Alsakhawi, Principal Investigator — Assistant Professor
Locations (1):
- Reham Alsakhawi, Giza, Egypt